CLINICAL TRIAL: NCT01986049
Title: Phase 3 Study Comparing Transversus Abdominis Plane Block After Caesarian Section Usin Bupivacaine 0.5% vs. Bupivacaine 0.25% vs. Placebo (Normal Saline).
Brief Title: Transversus Abdominis Plane (TAP) Block for Post Caesarian Pain
Acronym: TAPBlock
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: We never collected data or started to recruit participants
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Joel Yarmush, Anesthesiologist, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRBNet # 367320
Record Dates: First submitted 2013-11-07; First posted 2013-11-18 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2019-08

CONDITIONS: Obstetrical Complications From Sedation During Parturition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bupivicaine 0.5% (Experimental): Drug Bupivacaine 0.5%
  Interventions: Drug: Bupivicaine
- Bupivicaine 0.25% (Experimental): Drug Bupivacaine 0.25%
  Interventions: Drug: Bupivicaine
- Normal Saline (Placebo Comparator): Saline Normal
  Interventions: Drug: Bupivicaine

INTERVENTIONS:
Drug: Bupivicaine

SUMMARY:
Adding TAP block with Bupivacaine may decrease the use of PCA bolus use after caesarean section for pain relief.

DETAILED DESCRIPTION:
Participants in the study will be randomized to TAP block with 0.5% or 0.25% bupivacaine or with placebo (normal saline).

The number of PCA bolus used within 24 hours post cesarean section will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

Healthy pregnant (ASA II) patients presenting for planned Cesarean delivery at New York Methodist Hospital under combined spinal epidural anesthesia

Exclusion Criteria:

* They are unable or are unwilling to take part in the study
* They have a history of allergy to any of the medications to be used in the study
* They have a history of drug abuse or chronic pain or opioid use
* They weigh less than 60kg
* They have a multiple gestation, placental disease, preeclampsia other disease of pregnancy
* They have a contraindication to neuraxial anesthesia (i.e., bleeding problems, bacteremia, etc.)
* They are unable to understand instructions or questions related to the study
* ASA III or IV

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Transversus Abdominis Plane (TAP) Block for Post Caesarean Pain | The first post operative 24 hours
  In Patient Controlled analgesia (PCA) system, the patient receives a preset dose of morphine by pressing a button on a computerized pump that is connected to an IV catheter. With PCA the patient may receive a small continuous flow of morphine and add more morphine as needed to provide a more constant level of comfort. In this study, we will compare the number of PCAs used by the participants in each arm

SECONDARY OUTCOMES:
Decrease in the pain score as measured by Visual Analog Scale (VAS) | The first post operative 24 hours
  Visual Analog Scale (VAS) is a numeric scale to measure the pain intensity from 0 to 10, where 0 = no pain, (1-3) = mild pain, (4-6) = moderate pain, and (7-10) = severe pain. The worst imaginable pain = 10

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Weinberg, MD, Study Director — New York Methodist Hospital Hospital
Locations (1):
- New Yoyk Methodist Hospital, Brooklyn, New York, United States